CLINICAL TRIAL: NCT02389686
Title: Intra-operative Radiotherapy For Women With Ductal Carcinoma in Situ Breast Cancer After Nipple-sparing Mastectomy
Brief Title: Intra-operative Radiotherapy For Breast Cancer Women After NSM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liao Ning (Other)
Responsible Party: Sponsor-Investigator, Liao Ning, MD,PhD, Guangdong Academy of Medical Sciences
Organization: Guangdong Academy of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GGHBCRG-IORT-NSM
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Breast Neoplasms
Keywords: Ductal carcinoma in situ （DCIS）; Nipple-sparing mastectomy (NSM); Intraoperative radiotherapy (IORT); INTRABEAM
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Without Radiotherapy (No Intervention): Patients just accept nipple-sparing mastectomy (NSM) without radiotherapy.
- Intraoperative Radiotherapy (Experimental): Followed by nipple-sparing mastectomy (NSM),INTRABEAM IORT was carried out with a single dose of 16 Gy for nipple-areola complex (NAC).
  Interventions: Device: INTRABEAM (Carl Zeiss, Oberkochen, Germany)

INTERVENTIONS:
Device: INTRABEAM (Carl Zeiss, Oberkochen, Germany) — Boost with 16 Gy during NSM for nipple-areola complex (NAC)
  Arms: Intraoperative Radiotherapy

SUMMARY:
The role of NSM is still controversial, mainly because of concern about the oncologic safety of the nipple-areola complex (NAC).INTRABEAM (Carl Zeiss, Oberkochen, Germany) is the most widely used mobile intraoperative radiotherapy (IORT) device to date. This study aims to assess the value of the INTRABEAM system for breast cancer.

DETAILED DESCRIPTION:
Despite the advancement and increasing use of nipple-sparing mastectomy (NSM) is still carried out in a portion of breast cancer patients. However, the role of NSM is still controversial, mainly because of concern about the oncologic safety of the nipple-areola complex (NAC). Radiation therapy uses high-energy x-rays to damage tumor cells. Giving radiation during surgery followed by external-beam radiation to the entire breast may kill more tumor cells.INTRABEAM (Carl Zeiss, Oberkochen, Germany) is the most widely used mobile intraoperative radiotherapy (IORT) device to date. This study aims to broaden the application of the INTRABEAM system for breast cancer, investigating the feasibility of INTRABEAM IORT in NSM with breast reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Tumor diameter ≤3 cm
* Tumor from the papilla>2cm
* Low grade ductal carcinoma in situ
* Candidate for breast-conserving surgery
* Must have undergone lumpectomy with negative margins or minimal margin involvement
* Currently undergoing re-excision of the biopsy cavity and/or sentinel lymph node biopsy or axillary lymph node dissection
* No evidence of metastatic disease
* Informed consent

Exclusion Criteria:

* No informed consent
* Tumor size > 3 cm
* Tumor from the papilla≤2cm
* Intermediate or high grade ductal carcinoma in situ
* Invasive carcinoma
* No indication for a boost

Ages: 17 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2014-10; Primary Completion 2019-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Ipsilateral breast tumor recurrence rate after surgery within five years | Within 5 years after surgery
  Within 5 years after surgery,we should evaluate ipsilateral breast tumor recurrence and Disease free survival as the most important outcome measure

SECONDARY OUTCOMES:
Disease free survival after surgery within five years | Within 5 years after surgery
  Within 5 years after adjuvant chemotherapy,we should evaluateDisease free survival(DFS) rates as thet important outcome measure.
Overall survival after surgery within ten years | Within ten years after surgery
  After surgery,we should evaluate overall survival (OR)rates as the secondary important outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Liao Ning, MD,PhD, Study Director — Guangdong Academy of Medical Sciences
Locations (1):
- Guangdong Academy of Medical Sciences, Guangzhou, Guangdong, China